CLINICAL TRIAL: NCT06604754
Title: Effects of Virtual Reality Training on Balance and Fall Risk of Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of VR Training on Balance and Fall Risk of Patients With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Syeda Marium Nadeem
Record Dates: First submitted 2024-09-18; First posted 2024-09-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: COPD; VR; BBS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Based Training (Experimental): Virtual reality (VR) based balance training utilizes immersive digital environments to enhance balance and stability through interactive and engaging exercises. Patients wear VR headsets that create realistic scenarios where they perform various balance tasks, such as navigating virtual obstacles or maintaining stability on unstable surfaces. This technology offers the advantage of providing controlled, adjustable challenges that can be tailored to the patient's specific needs and progress. VR training often incorporates real-time feedback, which helps patients improve their balance in a motivating and dynamic setting.
  Interventions: Other: Assigned Intervention for VR Training
- Traditional Physical Therapy Based Training: (Active Comparator): Traditional physical therapy-based balance training focuses on improving stability and preventing falls through a variety of exercises and techniques. It typically begins with a comprehensive assessment to identify balance issues and set individualized goals. The training includes static exercises like single-leg stands, dynamic activities such as walking on uneven surfaces, and strengthening and flexibility exercises to enhance muscle control and range of motion. Coordination and functional training, including gait and daily activity simulation, are also integral. Additionally, patients receive education on fall prevention strategies and home safety. Regular monitoring ensures that the program is adjusted to the patient's progress and ongoing needs, ultimately enhancing balance and reducing fall risk.
  Interventions: Other: Assigned Intervention for Traditional Physical Therapy Training

INTERVENTIONS:
Other: Assigned Intervention for VR Training — In VR training patients use VR headsets to engage in virtual environments for 8 weeks where they perform exercises designed to enhance balance, coordination, and strength. Simultaneously, the VR platform incorporate pulmonary exercises that focus on improving breathing techniques, lung capacity, and overall respiratory health. Patients will engage in 3 sessions per week with total time duration of 45 to 60 minutes. VR-based training provides real-time feedback and adapts to the patient's progress, offering a comprehensive approach to rehabilitation that addresses both balance and pulmonary function in a motivating and controlled manner.
  Arms: Virtual Reality Based Training
Other: Assigned Intervention for Traditional Physical Therapy Training — In Traditional physical therapy balance training for patients with chronic obstructive pulmonary disease (COPD) involves exercises designed to improve stability, strength, and coordination for duration of 8 weeks. These exercises, such as static balance tasks, dynamic movement drills, and strength training, help address the balance deficits often seen in COPD patients due to muscle weakness and reduced physical activity. Additionally, pulmonary effects are managed through breathing exercises such as deep breathing and pursed lip breathing that enhance respiratory functions, improve lung capacity and efficiency.
  Arms: Traditional Physical Therapy Based Training:

SUMMARY:
The aim of this study is to determine whether Virtual Reality (VR) training has significant effects on balance and fall risk of patients with COPD, with a focus on the patient group (GOLD STANDARD I & II). Additionally, the study determines whether VR training is a reliable substitute for traditional physical therapy balance.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is the forth leading cause of mortality worldwide. COPD often impairs balance due to decreased physical activity, muscle weakness, and compromised respiratory function. Virtual Reality training addresses these issues by offering an immersive and engaging environment that enhances patient motivation and adherence to rehabilitation. The technology allows for personalized and controlled balance exercises, progressively increasing the difficulty to match the patient's skill level and providing real-time feedback. By integrating cognitive and motor tasks, VR promotes a comprehensive approach to balance training, improving sensory integration and postural control.

Research indicates that VR training can enhance both static and dynamic balance, helping patients maintain stability in various conditions. It improves the integration of sensory inputs crucial for balance, while also contributing to muscle strength and endurance. This results in a reduction in fall frequency, as patients become more adept at managing balance and are less likely to fall during daily activities. Additionally, VR training teaches specific fall prevention strategies and boosts patient confidence, which further mitigates the fear of falling-a common issue among COPD patients.

Incorporating VR training into physical therapy programs for COPD patients can be highly beneficial. Its ability to provide engaging and customizable exercises makes it a valuable tool in addressing balance issues and reducing fall risks. However, it is essential to ensure that VR training is conducted under proper supervision to avoid potential accidents, especially in patients with severe COPD or additional health concerns. Overall, VR training represents a significant advancement in rehabilitation, offering a novel and effective approach to managing balance and fall risks in COPD patients. The purpose of study is to determine whether VR training has significant effects on balance and fall risk of patients with COPD (GOLD standard stage I & II).

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Female
* Diagnosed with mild to moderate COPD (GOLD stages I-II)
* Age between 40-65 years
* BBS score above 35 will be included.
* COPD patients with oxygen saturation of above 88%.
* Patients able to follow instructions / commands.

Exclusion Criteria:

* Recent exacerbation of COPD requiring hospitalization within last 4 weeks.
* Diagnosed with severe cognitive impairments.
* Previous experience with VR-based rehabilitation.
* Use of medication that could affect exercise response.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Balance | 8 weeks
  Berg Balance Scale (BBS) is used to assess balance. It consists of a 14 item that evaluates a persons performance on particular functional task.
Functional Capacity | 8 weeks
  The Six Minute Walk Test (SMWT) is a widely used tool for assessing functional exercise capacity, especially in populations with pulmonary and cardiovascular conditions. The test is performed under controlled conditions with the patient encouraged to perform at their own pace and take breaks if needed. the distance covered is measured and any change in condition or symptoms are noted.
Peak Expiratory Flow rate | 8 weeks
  Peak expiratory flow rate (PEFR) Peak expiratory flow rate (PEFR) measured through digital spirometer. Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings
Forced Vital Capacity | 8 weeks
  Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal.
Forced Expiratory Volume in 1sec | 8 weeks
  Forced expiratory volume in 1sec (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal.
FVC/FEV1 ratio | 8 weeks
  The FVC/FEV1 ratio is crucial for differentiating between obstructive and restrictive lung patterns. It helps in diagnosing conditions like asthma and COPD, and in monitoring the progression or improvement of these diseases. In clinical practice, this ratio is used alongside other spirometric measurements and patient history to provide a comprehensive assessment of lung function.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No